CLINICAL TRIAL: NCT05740163
Title: Oral Immunotherapy for Egg Allergy in Children Aged 6 to 16
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: University of Oulu (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Rudiger Schultz, Specialist in Pediatric Allergology, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oral immunotherapy fo egg
Record Dates: First submitted 2023-01-16; First posted 2023-02-22 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Egg Allergy
Keywords: Oral immunotherapy; Egg allergy; Children
MeSH Terms: conditions — Egg Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Egg allergy with asthma with intervention (Experimental): Immunotherapy Egg product including egg white and yolk allergens
  Interventions: Dietary Supplement: Egg product including egg white and yolk allergens
- Egg allergy without asthma with intervention (Experimental): Immunotherapy Egg product including egg white and yolk allergens
  Interventions: Dietary Supplement: Egg product including egg white and yolk allergens
- Egg allergy with asthma without intervention (No Intervention): No intervention, control
- Egg allergy without asthma without intervention (No Intervention): No intervention, control

INTERVENTIONS:
Dietary Supplement: Egg product including egg white and yolk allergens — Egg product either meatball or bread roll or bun including egg white and yolk allergens delivered orally in increasing dosages daily.
  Arms: Egg allergy with asthma with intervention; Egg allergy without asthma with intervention

SUMMARY:
The aim of the study is to determine the efficacy of a 12-month egg oral immunotherapy (OIT) protocol with a cooked whole egg product including yolk and egg white.

Study hypothesis: With this method the risk for severe allergic reaction to egg protein is reduced and the diet can partly or completely be normalized.

DETAILED DESCRIPTION:
The prevalence of egg allergy among children varies from 0.5% to 3% and is thus the second most common food allergy in children. Until recently, the only treatment for egg allergy was in many cases a life-long avoidance of egg protein. Due to the large number of egg-allergic children, oral immunotherapy (OIT) to egg has been suggested to be of probable benefit to cure children with egg-allergy. Several studies have been conducted to evaluate the safety and clinical outcome of egg OIT. However, concerning efficacy and safety of egg OIT more data, and alternative procedures are required to gain a safe, simple and inexpensive immunotherapy protocol . Previous egg OIT studies have mainly used egg white in the immunotherapy, rather than more natural and inexpensive whole egg products.

The aim of this study is to determine the efficacy of a 12-month egg oral immunotherapy (OIT) protocol with a cooked whole egg product including yolk and egg white. Furthermore, the effects of whole egg OIT on humoral immune responses are investigated.

The investigators hypothesize that oral administration of a whole egg product with incremental dosing will increase the individual threshold for allergic reactivity to egg protein and may result in full tolerance without any reaction to egg.

Other study aims include investigating the differences in efficacy and side effects of whole-egg OIT in children with asthma and without asthma. In this study it is hypothesized that children with asthma have more symptoms than non-asthmatic children during the treatment. Furthemore, the level of asthma control during OIT is investigated.

The study is a prospective multicenter randomized open trial, investigating the efficacy, safety and immunological mechanisms of oral egg immunotherapy in children (aged 6 to 16). Children with egg allergy, egg avoidance diet, immediate reaction in a food challenge test for egg within the last six months and elevated serum egg-specific immunoglobulin E (IgE) levels, are recruited into the study. Children with uncontrolled asthma, severe cardiovascular disease and autoimmune disease or families with poor compliance are excluded from the study.

Study participants are divided into two groups: patients with asthma and without asthma. Both groups are separately randomized into immunotherapy or follow-up without the treatment. The immunotherapy and follow-up last 12 months in total. After 12 months of enrolment, participants in the follow-up group are entitled to take actively part in the egg OIT protocol.

In immunotherapy groups (asthma or no-asthma), meatball, bun or bread roll, including well-cooked whole-egg is given daily to the patients, starting from a minimal dosage (1/200 of the protein content of whole egg) and increasing the dosing every 1-2 weeks until a dosage of 1/5 of the protein content of a whole egg is reached. The initial dosage is given at the hospital outpatient clinic. The patients and their parents will be prepared for emergency treatment of severe allergic reactions and are given instructions to carry adequate medication with them. Patients in the intervention groups take levocetrizine 5 mg or cetirizine 10 mg daily until three months of maintenance dosage.

Blood samples, skin prick tests, lung function tests and exhaled nitric oxide levels are taken from all study participants. All the above-mentioned tests are taken before the therapy and at the time points of 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 16 years
* Elevated spesific serum IgE to egg (> 5 kU/l) and/or positive skin prick to egg allergen
* Positive oral food challenge for egg or anaphylaxis reaction to egg within the 6 months
* Diet free from egg in any form

Exclusion Criteria:

* Age less than 6 years or more than 16 years
* Poor asthma control or uncontrolled asthma
* Severe/significant cardiovascular disease
* Autoimmune disease
* Malignancy
* Medication: beta bloker, angiotensin-converting-enzyme inhibitors (ACE inhibitors), Monoamine oxidase inhibitors (MAOIs)
* Poor compliance
* Fear of immunotherapy
* Desensitization to alfa-gal-protein (mammalian meat allergy)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of oral egg immunotherapy | Within 12 months of study
  Total number of patients who achieved tolerance to egg protein during OIT (negative egg challenge) compared to the number of patients who received only partly tolerance or failed to develop any level of unresponsiveness.

SECONDARY OUTCOMES:
Safety of oral egg immunotherapy | Within 12 months of study
  Total number of participants with adverse events, and total number of adverse events evaluating the safety of our method
Specification of adverse reactions during egg OIT in patients without asthma | Within 12 months of study
  Subjective evaluation and grading of symptoms from different organ sides during OIT, using visual analogue score 0-10 (VAS) in patients without asthma
Number and severity of anaphylactic reactions during OIT without asthma | Within 12 months of study
  Number and severity of anaphylaxis during OIT (Grading of anaphylaxis using Samsons criteria, grade1-5) in patients without asthma
Specification of adverse reactions during OIT in patients with asthma | Within 12 months of study
  Subjective evaluation and grading of symptoms from different organ sides during OIT, using visual analogue score 0-10 (VAS) in patients with asthma
Number and severity of anaphylactic reactions durin OIT in patients with asthma | Within 12 months of study
  Number and severity of anaphylaxis in patients with asthma (Grading of anaphylaxis using Samsons criteria, grade 1-5) in patients with asthma.
Effect of immunotherapy on the level of whole serum IgE | Within 12 months of study
  Changing values in blood samples during OIT describing changes in whole IgE by determining values before OIT and after 6 and 12 months of OIT.
Effect of immunotherapy on the level of specific egg IgE (sIgE) | Within 12 months of study
  Changing values in blood samples during OIT describing changes in egg sIGE by determining values before OIT and after 6 and 12 months of OIT.
Effect of immunotherapy on white blood cells | Within 12 months of study
  Changing values in blood samples during OIT describing changes in the white blood-cell count by determining values before OIT and after 6 and 12 months of OIT.
Effect of immunotherapy on the level of egg IgG4 (sIgG4) | Within 12 months of study
  Changing values in blood samples during OIT describing changes in the egg sIgG4 by determining values before OIT and after 6 and 12 months of OIT.
Effect of immunotherpay on heat stable, egg components | Within 12 months of study
  Changing values in blood samples during OIT describing changes in the heat stable molecules of Gal d1 and Gal d2 by determining values before OIT and after 6 and 12 months of OIT.
Effect of immunotherpay on the activity of eosinophils | Within 12 months of study
  Changing values in blood samples during OIT describing changes in the level of eosinophilic cationic protein (ECP) by determining values before OIT and after 6 and 12 months of OIT.
Changes in parameters describing lung inflammation in patients with asthma | Within 12 months of study
  Comparison of values of exhaled nitric oxide (ppb) and serum ECP (ug/l) by comparing the results 6 and 12 months after starting OIT to baseline values before OIT.
Changes in parameters describing lung inflammation in patients without asthma | Within 12 months of study
  Comparison of values of exhaled nitric oxide (ppb) and serum ECP (ug/l) by comparing the results 6 and 12 months after starting OIT to baseline values before OIT.
Changes in lung function parameters during OIT in patients with asthma and > 7 years of age | Within 12 months of study
  Effect of OIT on parameters describing lung function in children over > 7 years of age employing flow-volume spirometry. Changing levels of FEV1 (l) and PEF (l/s) will be recorded.
Changes in lung function parameters during OIT in patients with asthma < 7 years of age | Within 12 months of study
  Effect of OIT on parameters describing lung function in children < 7 years of age employing impedance oscillometry. Changing levels of 5Hz resistance (R5, kPa/l/s) and total impedance (Z5, kPa/l/s) will be recorded.
Changes in lung function parameters during OIT in patients without asthma and > 7 years of age | Within 12 months of study
  Effect of OIT on parameters describing lung function in children over > 7 years of age and without ashma employing flow-volume spirometry. Changing levels of FEV1 (l) and PEF (l/s) will be recorded.
Changes in lung function parameters during OIT in patients without asthma and < 7 years of age | Within 12 months of study
  Effect of OIT on parameters describing lung function in children < 7 years of age and without asthma employing impedance oscillometry. Changing levels of 5Hz resistance (R5, kPa/l/s) and total impedance (Z5, kPa/l/s) will be recorded.
Recording of asthma symptoms during egg OIT in patients with asthma | Within 12 months of study
  Subjective evaluation and grading of asthmatic symptoms during OIT, using visual analogue score (VAS).
Recording of asthma symptoms during egg OIT in patients without asthma | Within 12 months of study
  Subjective evaluation and grading of asthmatic symptoms during OIT, using visual analogue score (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger Schultz, MD., PhD, Principal Investigator — Tampere University Hospital
Locations (2):
- Finland (2):
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No